CLINICAL TRIAL: NCT00503711
Title: An Open Label, Phase I, Rising Multiple Dose, Single Centre Study to Determine the PK and Tolerability of ZD6474 at Different Dose Levels in Chinese Patients With Solid Malignancy Tumor
Brief Title: Phase I Chinese PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4200L00004
Record Dates: First submitted 2007-07-18; First posted 2007-07-19 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Advanced Solid, Malignant Tumors
Keywords: ZD6474 PK
MeSH Terms: conditions — Neoplasms | interventions — vandetanib

ARMS (3):
- 100 mg Vandetanib eod (Experimental): 100 mg Vandetanib every other day dosing
  Interventions: Drug: Vandetanib
- 100 mg Vandetanib od (Experimental): 100 mg Vandetanib once daily dosing
  Interventions: Drug: Vandetanib
- 300 mg Vandetanib od (Experimental): 300 mg Vandetanib once daily dosing
  Interventions: Drug: Vandetanib 300 mg

INTERVENTIONS:
Drug: Vandetanib — 100 mg every other day, 100mg once daily
  Other Names: ZD6474; ZACTIMA™
  Arms: 100 mg Vandetanib eod; 100 mg Vandetanib od
Drug: Vandetanib 300 mg — 300mg once daily
  Other Names: ZD6474; ZACTIMA™
  Arms: 300 mg Vandetanib od

SUMMARY:
An open, phase 1 to assess the PK of rising doses of ZD6474 when administered daily in Chinese patients with advanced solid malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

* histological and/or cytological confirmation of a malignant solid tumor
* refractory to standard therapies or for which no appropriate therapies exist
* WHO performance status 0-2

Exclusion Criteria:

* patients with brain tumors or symptomatic cerebral metastases
* systemic anticancer therapy within the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-09; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) (0-24) (ng.h/mL) after single dose | Blood sample is collected at 1, 2, 4, 6, 8, 10 & 24 hour after first single dose on day 1

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Research Site, Guangzhou, China

REFERENCES:
- [Background] Zhang L, Li S, Zhang Y, Zhan J, Zou BY, Smith R, Martin PD, Jiang Y, Liao H, Guan Z. Pharmacokinetics and tolerability of vandetanib in Chinese patients with solid, malignant tumors: an open-label, phase I, rising multiple-dose study. Clin Ther. 2011 Mar;33(3):315-27. doi: 10.1016/j.clinthera.2011.04.005. PMID 21600385